CLINICAL TRIAL: NCT03788577
Title: Impact of Oligonol to Cardiometabolic Risk and Muscular Health: a Randomized Controlled Trial
Brief Title: Impact of Oligonol to Cardiometabolic Risk and Muscular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2018-05-004B
Record Dates: First submitted 2018-12-19; First posted 2018-12-27 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2020-02

CONDITIONS: Muscle Loss; Muscle Weakness; Quality of Life
MeSH Terms: conditions — Muscular Atrophy; Muscle Weakness

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oligonol intake group (Experimental): This experimental arm will be applied for Oligonol 200mg/tab 1 tab per day. The program will last for 12 weeks.
  Interventions: Dietary Supplement: Oligonol intake
- Placebo group (Placebo Comparator): This Placebo arm will be given capsules made of starch 1 tab per day. The program will last for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oligonol intake — Major intervention of Oligonol component , as suggested Oligonol safe dose for adults is 200mg per day.
  Arms: Oligonol intake group
Dietary Supplement: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
This project will mainly focus on Middle and old-aged adults, and examine whether Cardiovascular and metabolic risks can be reduced. In the meanwhile, this project will develop strategies for improving muscle loss , muscle strength decline, and the quality life of the elderly.

DETAILED DESCRIPTION:
Cardiovascular diseases are common among the elder. However, previous researches mainly focus on observational research or small scale clinical trial, and the subjects are mainly youth. Therefore, this project hope to understand whether Oligonol can reduce Cardiovascular and metabolic risks among senior adults. Consequently,improve muscle loss muscle strength decline, quality of old adults life. This project design may potentially develop new strategies for curing Sarcopenia as well.

ELIGIBILITY:
Inclusion Criteria:

* People who aged more than 50 years
* Patients with following characteristics:
* feeling loss in activity.
* detecting decline in self's walking speed.
* feeling tired of doing everything.
* having fallen down last year.
* People can accept undergoing MRI
* People willing to follow the program and cooperate with us for following tracking.
* People who are neither vegan nor vegetarian

Exclusion Criteria:

* Walking speed less than 0.3m/s
* People with any disease affecting their limbs, including:
* having fracture on limbs in the past 6 months.
* having severe arthritis in the past 6 months
* any other whom PI recognized as weak control of their nervous system( e.g.: Parkinson's disease and stroke).
* People with intermittent limp caused by peripheral artery diseases
* People with weak control of mental disorder
* People with weak control of Cardiopulmonary disease
* People with weak control of Malignant tumor
* People with weak control of kidney diseases (GFR < 30 mL/min/1.73 m2 for at least 3 months)
* People with visual impairment and hearing disorder who cannot complete the program.
* People who are unable to undertake MRI
* Any other condition that PI recognized as not suitable.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Changes from baseline muscle after 12 weeks | baseline,12 weeks
  Change from baseline muscle via MRI after 12 weeks.
Changes from baseline fat content of leg after 12 weeks | baseline,12 weeks
  Change from baseline fat content of leg via MRI after 12 weeks.
Changes form baseline chair-stand after 12 weeks | baseline, 12 weeks
  measured by the time of chair-stand after 12 weeks.
Changes form baseline muscle strength after 12 weeks | baseline, 12 weeks
  measured by hand grip distance after 12 weeks.
Change from baseline Nutrition intake after 12 weeks | baseline, 12 weeks
  measured by Mini-nutritional assessment questionnaire. ranged 0-30, higher values represent a better condition
Change from baseline depression after 12 weeks | baseline, 12 weeks
  measured by the Center for Epidemiological Studies-Depression (CES-D) ranged 0-60, higher values represent a worse condition
Change from baseline endurance after 12 weeks | baseline, 12 weeks
  measured by 6-minute walk distance
Change from baseline walking speed after 12 weeks | baseline, 12 weeks
  measured by six-meter walking speed
Change from baseline timed up and go test after 12 weeks | baseline, 12 weeks
  measured by timed up and go test (TUG)

SECONDARY OUTCOMES:
Change from baseline numbers of Complete blood count after 12 weeks | baseline,12 weeks
  Change from baseline numbers of Complete blood count after 12 weeks
Change from baseline concentration of Albumin after 12 weeks | baseline,12 weeks
  Change from baseline concentration of Albumin after 12 weeks
Change from baseline concentration of Alanine Aminotransferase (ALT) after 12 weeks. | baseline,12 weeks
  Change from baseline concentration of Alanine Aminotransferase (ALT) after 12 weeks.
Change from baseline concentration of Aspartate Aminotransferase (AST) after 12 weeks. | baseline,12 weeks
  Change from baseline concentration of Aspartate Aminotransferase (AST) after 12 weeks.
Change from baseline concentration of blood urea nitrogen after 12 weeks | baseline,12 weeks
  Change from baseline concentration of blood urea nitrogen after 12 weeks
Change from baseline concentration of Creatinin after 12 weeks | baseline,12 weeks
  Change from baseline concentration of Creatinin after 12 weeks
Change from baseline concentration of Fasting glucose after 12 weeks | baseline,12 weeks
  Change from baseline concentration of Fasting glucose after 12 weeks
Change from baseline concentration of Total Cholesterol after 12 weeks | baseline,12 weeks
  Change from baseline concentration of Total Cholesterol after 12 weeks
Change from baseline concentration of Triglyceride after 12 weeks | baseline,12 weeks
  Change from baseline concentration of Triglyceride after 12 weeks
Change from baseline concentration of high-density lipoprotein cholesterol after 12 weeks | baseline,12 weeks
  Change from baseline concentration of high-density lipoprotein cholesterol after 12 weeks
Change from baseline concentration of low-density lipoprotein cholesterol after 12 weeks | baseline,12 weeks
  Change from baseline concentration of low-density lipoprotein cholesterol after 12 weeks
Change from baseline concentration of high-sensitivity C-reactive protein after 12 weeks | baseline,12 weeks
  Change from baseline concentration of high-sensitivity C-reactive protein after 12 weeks
Change from baseline concentration of dehydroepiandrosterone after 12 weeks | baseline,12 weeks
  Change from baseline concentration of dehydroepiandrosterone after 12 weeks
Change from baseline concentration of 25-(OH)-Vit. D after 12 weeks | baseline,12 weeks
  Change from baseline concentration of 25-(OH)-Vit. D after 12 weeks
Change from baseline concentration of Leptin after 12 weeks | baseline,12 weeks
  Change from baseline concentration of 25-(OH)-Vit. D after 12 weeks
Change from baseline concentration of urine protein after 12 weeks | baseline,12 weeks
  Change from baseline concentration of urine protein after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Kung Chen, MD.PhD., Principal Investigator — Center for Healthy Longevity and Aging Sciences, National Yang Ming University
Locations (1):
- Taipei Veteran General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No